CLINICAL TRIAL: NCT02397837
Title: Pramipexole in Bipolar Disorder: Targeting Cognition (PRAM-BD)
Brief Title: Targeting Cognition in Bipolar Disorder With Pramipexole
Acronym: PRAM-BD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Zucker Hillside Hospital (Other); Northwell Health (Other); National Institute of Mental Health (NIMH) (NIH); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Katherine Burdick, Lead Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017P001185; 1R01MH102257 (NIH); 1R01MH102309 (NIH)
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Cognition
MeSH Terms: conditions — Bipolar Disorder | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pramipexole (Experimental): Pramipexole, by mouth. Dosing will be initiated at 0.25 mg on night one, followed by 0.25 mg twice-a-day day two onward, and increased every week to a target of 4.5 mg/day for the 12-week duration of the study.
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Placebo, by mouth. Dosing will be initiated at 0.25 mg on night one, followed by 0.25 mg twice-a-day day two onward, and increased every week to a target of 4.5 mg/day for the 12-week duration of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole — Up to 4.5mg, PO, (by mouth) per day of the 12-week study.
  Other Names: Mirapex
  Arms: Pramipexole
Drug: Placebo — placebo match study drug
  Arms: Placebo

SUMMARY:
Converging evidence suggests that patients with bipolar disorder suffer from deficits in neurocognitive functioning that persist, despite remission of acute affective symptoms. These impairments contribute directly to functional disability, highlighting the need for interventions above and beyond standard treatments in order to achieve a full inter-episode recovery. The current study aims to investigate the safety and efficacy of a dopamine agonist (pramipexole), on these persistent cognitive abnormalities in euthymic bipolar patients using a placebo-controlled, adjunctive, 12-week trial design.

DETAILED DESCRIPTION:
All eligible participants will undergo study visits at screening, baseline (week 0), week 1, week 2, week 3, week 4, week 6, week 8, and week 12, (end of study).

Randomization will be conducted via a computer generated program and all study staff will be blinded unless un-blinding is required for safety reasons. Subjects will be randomized on a 1:1 ratio with stratification for concomitant antipsychotic status and depression at baseline (HRSD <8 vs > 8). Study drug will be blinded and matched to placebo. Adapting from our previous work in BD and according to package labeling, the dosage titration schedule will be slow and flexible. Dosing will be initiated at 0.25 mg QHS on night one, followed by 0.25 mg BID day two onward, and increased every week to a target of 4.5 mg/day. As compared with our previous maximum 1.5 mg/day (Burdick et al. 2012), we opted to allow up to 4.5 mg/day (the maximum approved dosage in Parkinson's disease) to ensure adequate target engagement. We are familiar with this dose range, as 4.5 mg/day was allowed in our study in BD depression (Goldberg et al. 2004). Dosing will be flexible based on side effects; however, if 1.5 mg/day cannot be tolerated, the subject will be discontinued. Titration will occur up to week 6 and then efforts will be made to maintain the same dose until the completion of the trial (week 12).

ELIGIBILITY:
Inclusion criteria:

* Age 18-65
* DSM-IV BD I or II diagnosis
* Affective stability, defined by a Young Mania Rating Scale (YMRS) rating of < 8 and a Hamilton Depression Rating Scale (HRSD) rating of < 16 at screening and baseline. We will further require that any subsyndromal depression has not significantly worsened in the 4 weeks prior to randomization so as to avoid enrolling subjects who are on the verge of a full depressive episode.
* Evidence of clinically-significant neurocognitive impairment at screening
* Clinically-acceptable, stably-dosed, mood stabilizing medication regimen for > 1 month prior to enrollment, with no medication changes planned over the 12-week study period.

Exclusion Criteria:

* History of CNS trauma, neurological disorder, ADHD, or learning disability
* Positive urine toxicology or DSM-IV diagnosis of substance abuse/dependence within 3 months
* Active, unstable medical problem that may interfere with cognition
* Recent history of rapid-cycling
* Abnormal lab or ECG result at screen
* History of heart failure
* Significant suicidal risk (HRSD item 3 > 2 or by clinical judgment)
* Estimated IQ in MR range as per Wide Range Achievement Test (WRAT) standard score of less than 70
* Pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (including oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
* Women who are breastfeeding
* Participation in any other investigational cognitive enhancement study within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Burdick, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Anil Malhotra, MD, Principal Investigator — The Zucker Hillside Hospital, North Shore LIJ- Health System
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] Burdick KE, Braga RJ, Nnadi CU, Shaya Y, Stearns WH, Malhotra AK. Placebo-controlled adjunctive trial of pramipexole in patients with bipolar disorder: targeting cognitive dysfunction. J Clin Psychiatry. 2012 Jan;73(1):103-12. doi: 10.4088/JCP.11m07299. Epub 2011 Nov 29. PMID 22152405
- [Background] Goldberg JF, Burdick KE, Endick CJ. Preliminary randomized, double-blind, placebo-controlled trial of pramipexole added to mood stabilizers for treatment-resistant bipolar depression. Am J Psychiatry. 2004 Mar;161(3):564-6. doi: 10.1176/appi.ajp.161.3.564. PMID 14992985

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol enrollment of 103 is the total number of participants who signed a consent form. 63 were randomized to a treatment group. The discrepancy between 103 and 63 is the total number of participants who completed a screen visit but failed to randomize (N=40).
Period: Overall Study
Arm/Group | Pramipexole | Placebo
Started | 33 | 30
Completed | 26 | 24
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole | Placebo | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 30 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 14 | 21
  White | 19 | 14 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 30 | 63

OUTCOME MEASURES:

1. Primary Outcome: MATRICS Consensus Cognitive Battery
Description: MATRICS Consensus Cognitive Battery (MCCB) as measure of Neurocognitive/Functional Measures is a standardized battery designed to measure cognitive functioning in people with schizophrenia. The MCCB is represented as a composite T score. This T-score scale has a mean of 50 and a standard deviation of 10, where higher scores reflect better performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 33 | 30
T-score | 35.45 (12.33) | 38.07 (10.45)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.38, t-test, 2 sided

2. Primary Outcome: MATRICS Consensus Cognitive Battery
Description: as for outcome 1
Time Frame: Week 6
Population: The discrepancy in participants analyzed here compared to baseline is due to an early termination from study of 5 participants in pramipexole group and 4 participants in placebo group.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 28 | 26
T-score | 35.57 (13.87) | 39.81 (11.01)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.22, t-test, 2 sided

3. Primary Outcome: MATRICS Consensus Cognitive Battery
Description: as for outcome 1
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 26 | 24
T-score | 36.46 (13.61) | 41.50 (11.47)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.17, t-test, 2 sided

4. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: Mean change of symptoms of mania throughout the study. YMRS contains 7 items rated from 0 (symptom absent) to 4 (severe symptom) and 4 items scored 0 (symptom absent) to 8 (severe symptom), with total range from 0 to 60, where higher score indicates manic symptoms.
Time Frame: Baseline and week 12
Population: Average change in YMRS based on baseline and week 12 score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 33 | 30
score on a scale | -0.92 (2.21) | -0.57 (1.88)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.55, t-test, 2 sided

5. Secondary Outcome: Hamilton Rating Scale for Depression (HRSD)
Description: Mean change of symptoms of depression throughout the study. HRSD consists of 14 items, each defined by a series of symptoms. Each item is rated on a 5-point scale, ranging from 0 (not present) to 4 (severe), with a total score range of 0-56, where higher score indicates more depressive symptoms.
Time Frame: Baseline and week 12
Population: Average change in HRSD based on baseline and week 12 score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 33 | 30
score on a scale | -0.24 (3.78) | -.22 (3.66)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.99, t-test, 2 sided

6. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: Mean change for positive symptoms throughout the study. BPRS consists of 18 items, each defined by a series of symptoms. Each item is rated on a 7-point scale, ranging from 1 (not observed) to 7 (very severe), with a total score range from 18-126, where higher scores indicate psychiatric symptoms.
Time Frame: Baseline and week 12
Population: Average change in BPRS based on baseline and week 12 score.The discrepancy in participants analyzed here compared to participant flow is due to available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 32 | 29
score on a scale | -0.63 (3.53) | -0.61 (3.70)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.98, t-test, 2 sided

7. Secondary Outcome: Number of Participants With Suicidal Acknowledgements
Description: Number of individual participants who acknowledged at least one item on the Columbia Suicide Severity Rating Scale (C-SSRS) over the 12-week study period. Examples of items on the scale are suicidal ideation (having thoughts, planning) and suicidal behavior (preparing, attempting).
Time Frame: up to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 33 | 30
Participants | 0 | 5
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; Tabulation of participants with suicidal acknowledgements over 12-week study

8. Secondary Outcome: The Probabilistic Stimulus Selection Task
Description: The probabilistic selection task assesses the tendency to learn from positive versus negative outcomes. In the probabilistic stimulus selection task, participants are trained to choose one of two paired stimuli; three sets of paired stimuli are shown in total (AB, CD, and EF) and are presented randomly during the training period. To minimize verbal encoding, stimuli are Japanese Hiragana characters. Probabilistic feedback regarding the "correct" choice is provided. We report the mean percentage of accuracy on choosing the correct paired stimuli among the two treatment groups.
Time Frame: Baseline
Population: The discrepancy in participants analyzed from participants in Participant Flow is due to availability of data because of software issues in running task.
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 18 | 21
percentage of accuracy | 56.94 (17.00) | 67.56 (20.12)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.09, t-test, 2 sided

9. Secondary Outcome: The Probabilistic Stimulus Selection Task
Description: as for outcome 8
Time Frame: Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 19 | 18
percentage of accuracy | 56.91 (22.60) | 56.94 (22.67)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 1.00, t-test, 2 sided

10. Secondary Outcome: The Probabilistic Stimulus Selection Task
Description: as for outcome 8
Time Frame: Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Pramipexole | Placebo
Number analyzed (Participants) | 19 | 19
percentage of accuracy | 59.54 (21.59) | 50.99 (16.04)
Statistical Analysis 1: Comparison: Pramipexole vs Placebo; Test type: Other; p = 0.17, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data collected from time of randomization/baseline visit through week 12 visit (end of study).
Arm/Group | Pramipexole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 18/33 | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramipexole (N=33) | Placebo (N=30)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Poor Coordination (General disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Ringing in Ears (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Painful Urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Menstrual Irregularity (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Difficulty Sleeping (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Poor Concentration (General disorders) | 2 (2) | 0 (0)
General malaise (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Decreased Energy (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Zucker Hillside Hospital Site (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT02397837/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Brigham and Women's Hospital Site (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT02397837/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT02397837/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan: Mount Sinai School of Medicine Site (2017-05-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT02397837/Prot_SAP_003.pdf